CLINICAL TRIAL: NCT02201576
Title: Treatment of Chronic Active Antibody-mediated Rejection With Bortezomib in Kidney Transplantation
Brief Title: Bortezomib in Rejection of Kidney Transplants
Acronym: TRIBUTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Fondation Centaure (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P120119
Record Dates: First submitted 2014-07-17; First posted 2014-07-28 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2019-10

CONDITIONS: Chronic Antibody-mediated Transplant Rejection
Keywords: Chronic antibody-mediated rejection,; transplant rejection, kidney transplantation,; proteasome inhibitor,; anti-HLA antibodies,; immunosuppressive agents
MeSH Terms: interventions — Bortezomib; Plasma Exchange; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bortezomib (Experimental): Five plasma exchanges, two cycles of bortezomib + dexamethasone, 4 courses of polyclonal intravenous immunoglobulins
  Interventions: Drug: Bortezomib
- Control (Active Comparator): Five plasma exchanges, dexamethasone, 4 courses of polyclonal intravenous immunoglobulins
  Interventions: Drug: Plasma exchanges and intravenous immunoglobulins

INTERVENTIONS:
Drug: Bortezomib — 1. Five plasma exchanges +0.1 g/kg of intravenous immunoglobulins at the end of each course
  2. two cycles of bortezomib (1.3 mg/m2 IV at day-1, day-4, day-8, day-11) + oral dexamethasone (20 mg po at day-1, day-4, day-8, day-11)
  3. four courses of polyclonal intravenous immunoglobulins every three weeks (2g/kg, the first two courses are performed simultaneously with the two bortezomib cycles)
  Other Names: Velcade
  Arms: Bortezomib
Drug: Plasma exchanges and intravenous immunoglobulins — 1. Five plasma exchanges +0.1 g/kg of intravenous immunoglobulins at the end of each course
  2. four courses of polyclonal intravenous immunoglobulins every three weeks (2g/kg)
  3. oral dexamethasone (20 mg po at day-1, day-3, day-5, day-7 of the two first intravenous immunoglobulins courses)
  Arms: Control

SUMMARY:
The purpose of the study is to assess the efficacy of bortezomib, in association with steroids, plasma exchange, and polyclonal intravenous immunoglobulins, in the treatment of chronic antibody mediated rejection due to donor specific anti-HLA antibodies, in kidney transplant recipients

DETAILED DESCRIPTION:
Chronic active antibody-mediated rejection (AMR) is considered as a main cause of late allograft losses in kidney transplant recipients. It is due to the occurrence of de novo donor-specific anti-HLA antibodies (DSA), i.e. antibodies synthetized by the recipient after transplantation against its transplant. There is currently to efficient treatment. The purpose of our study is to determine the efficacy of bortezomib, a proteasome inhibitor, in the treatment of chronic active antibody-mediated rejection, in association with steroids, plasma exchanges, and polyclonal intravenous immunoglobulins. Patients are recipients of a first or a second kidney transplant for more than 3 months. They display de novo DSA i.e. DSA not detected the day of transplantation and in pre-transplant sera.. They display signs of chronic active AMR on kidney biopsy i.e. a glomerulitis (g) + peritubular capillaritis (ptc) Banff score g+ptc ≥ 2, with or without severe chronic glomerulopathy (Banff score cg<3). Kidney biopsy may have been performed systematically or because of: :

1. detection of de novo DSA ,
2. and /or proteinuria (> 0.5 g/24h)
3. and /or slow graft dysfunction protocol biopsy Primary endpoint is a combined endpoint one year after inclusion, consisting of the stabilization of histological lesions on a new kidney biopsy (delta g+ptc ≤1 and delta cg < 1) and a decrease in DSA mean fluorescence intensity > 50%.

ELIGIBILITY:
Inclusion Criteria:

* recipients of a first or a second kidney transplant for more than 3 months
* age over 18 years
* with de novo donor specific antibodies (DSA), i.e. antibodies not detected the day of transplantation and in pre-transplant sera
* with histological lesions of chronic active antibody-mediated rejection (glomerulitis + peritubular capillaritis banff score and chronic glomerulopathy (g+ptc ≥ 2) on a graft biopsy performed because of renal function deterioration, proteinuria, detection of de novo DSA, or on a systematic biopsy
* written informed consent
* Given the teratogenic risks described in the SPCs of Velcade and Cellcept:

  * Women of child bearing age must have a negative pregnancy test the day of the inclusion and should use at least one effective contraceptive method before start of medication during the treatment and during the study
  * Men old enough to procreate have to use condoms during the treatment and at least 90 days after the last intake of the treatment during the study. Moreover, given SPCs of Cellcept, it is recommended that female partners to use an effective method of contraception treatment and for 90 days after the last mycophenolate intake by the partner male
* affiliated with social security health insurance
* patients with cell rejection lesions associated with chronic humoral rejection lesions active may be included in the study. This rejection can be treated with 3 boluses of 500 mg of methyl prednisolone prior to inclusion.

Exclusion Criteria:

* patient with preformed DSA
* recipient of a 3rd or 4th kidney transplant
* recipient of a transplant combined with another not renal organ
* patient with a history of humoral acute rejection during the current transplantation
* estimated GFR below 20 ml/min/1,73m2
* severe transplant glomerulopathy (cg score = 3)
* severe peripheral neuropathy, thrombopenia < 100 000 mm3 , neutropenia < 1000 mm3 and/or an uncontrolled evolutionary infection
* chronic active hepatitis B (positive HBs antigen or HBV DNA), positive chronic hepatitis C and/or known HIV infection
* allergy to bore or bortezomib or to one of the excipient
* hepatic failure, abnormal liver tests (bilirubin >3N, transaminases >3n), infiltrative pneumopathy, pericarditis
* risk of non-adherence to treatment or protocol
* inclusion in another clinical therapeutic trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-02-11 (Actual); Primary Completion 2020-07-16 (Actual); Study Completion 2020-07-16 (Actual)

PRIMARY OUTCOMES:
histological lesions of humoral rejection and immunodominant donor specific antibody | one year
  Between inclusion biopsy and end of study biopsy delta g+ptc ≤1 and delta cg < 1 (Banff score of glomerulitis (g) capillaritis (ptc) and chronic allograft glomerulopathy (cg) Between inclusion and end of study, decrease in mean fluorescence intensity (MFI) of the immunodominant donor specific anti-HLA antibody (DSA with the highest MFI) by Luminex greater than 50%

SECONDARY OUTCOMES:
histological lesions of humoral rejection | one year
  Between inclusion biopsy and end of study biopsy delta g+ptc ≤1 and delta cg < 1 (Banff score of glomerulitis (g) capillaritis (ptc) and chronic allograft glomerulopathy (cg)
immunodominant donor specific antibody | one year
  Between inclusion and end of study, decrease in mean fluorescence intensity (MFI) of the immunodominant donor specific anti-HLA antibody (DSA with the highest MFI) by Luminex greater than 50%
all donor specific antibodies at one year | one year
  Between inclusion and end of study, variation of the title of each DSA and the sum of the DSAs
all donor specific antibodies | 6 months
  Between inclusion and month-6, evolution in mean fluorescence intensity (MFI) of all donor specific anti-HLA antibodies by Luminex
Histological lesions | one year
  Description of all histological lesions observed at one-year biopsy according to the Banff classification and comparison with inclusion biopsy: acute cellular rejection, interstitial fibrosis and tubular atrophy, chronic vascular lesions (arteriolar hyalinosis, fibro-intimal thickening), chronic rejection (transplant glomerulopathy, fibroproliferative endarteritis)
renal function and proteinuria | one year
  Evolution between inclusion and end of study at one-year of serum creatinine, estimated GFR (MDRD formula), proteinuria output, proteinuria/creatinuria ratio
Safety of bortezomib in renal transplant recipients | one year
  Infectious and non-infectious adverse events occurring during study in the two arms of treatment
Patient and graft survival | one year
T and B lymphocytes subsets with bortezomib | one year
  Flow cytometry study of T and B lymphocytes subsets at inclusion, month-6 and month-12 in patients treated with bortezomib

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Legendre, MD, PhD, Study Chair — Assistance Publique - Hôpitaux de Paris; Renaud Snanoudj, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Necker Enfants-malades, Paris, France